CLINICAL TRIAL: NCT02484378
Title: CER-001 Atherosclerosis Regression ACS Trial; A Phase II Multi-Center, Double-Blind, Placebo-Controlled, Dose-Focusing Trial Of Cer-001 In Subjects With Acute Coronary Syndrome
Brief Title: CER-001 Atherosclerosis Regression ACS Trial
Acronym: CARAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cerenis Therapeutics, SA (Industry)
Collaborators: South Australian Health and Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CER-001-CLIN-010
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2017-01

CONDITIONS: Acute Coronary Syndromes
Keywords: ACS; IVUS; HDL
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — CER-001

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CER-001 (Experimental): CER-001 infusion
  Interventions: Drug: CER-001
- Placebo (Placebo Comparator): Placebo infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CER-001 — Engineered pre-beta HDL particle
  Other Names: CAS 1383435-67-3
  Arms: CER-001
Drug: Placebo — Normal saline
  Other Names: Placebo for CER-001
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the impact of ten intravenous infusions of 3 mg/kg CER 001 vs. placebo, given at weekly intervals for ten weeks, on atherosclerotic plaque volume as measured by coronary IVUS, when administered to subjects presenting with Acute Coronary Syndrome (ACS) with significant plaque volume.

DETAILED DESCRIPTION:
Subjects will be required to have at least one epicardial coronary artery suitable for IVUS imaging. A suitable target artery for IVUS imaging will be determined at baseline as having stenosis of up to 50% and meeting all angiographic inclusion criteria. Subjects having met all eligibility criteria will be randomized to receive an intravenous infusion of CER 001 (3 mg/kg) or placebo within 14 days of event presentation. Randomized subjects will then return at 7 day intervals for nine additional infusions. A follow up IVUS will be conducted at 14 days after the last infusion. The total study duration from randomization to follow up IVUS for a completed study can range from approximately 9 to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female greater than 18 years of age
* Acute coronary syndrome (myocardial infarction or unstable agina)
* Angiographic evidence of coronary artery disease with suitable "target" coronary artery for IVUS evaluation

Exclusion Criteria:

* Females of child-bearing potential
* Angiographic evidence of >50% stenosis of the left main artery
* Uncontrolled diabetes (HbA1C>10%)
* Hypertriglyceridemia (>500 mg/dL)
* Congestive heart failure (NYHA class III or IV)
* Ejection fraction <35%
* Uncontrolled hypertension (SBP >180 mm Hg)
* Known major hematologic, renal, hepatic, metabolic, gastrointestinal or endocrine dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Nominal Change in Percent Atheroma Volume (PAV) | Baseline to 12 weeks
  The nominal change from baseline to follow-up (at 12 weeks) in the percent atheroma volume (PAV) in the target coronary artery assessed by 3 dimensional (3D) IVUS

SECONDARY OUTCOMES:
Nominal Change in Normalized Total Atheroma Volume (TAV) | Baseline to 12 weeks

OTHER OUTCOMES:
Major Cardiovascular Events (MACE) | 12 weeks
  Episodes of all death, non-fatal myocardial infarction, resuscitated cardiac arrest, non-fatal stroke, fatal stroke, coronary revascularization procedures [percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG)], hospitalization for unstable angina, urgent visit or hospitalization for congestive heart failure (CHF), any admission for a procedure for the treatment of PVD (including cerebrovascular procedures) and urgent readmission with chest pain. The events will be reviewed and adjudicated by the Clinical Endpoint Committee according to established definitions. This study is not powered for MACE endpoints.
Lipid Profiles | Throughout the 12 week study period
  Pre-dose lipid profiles, including low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C), total cholesterol (TC), unesterified cholesterol (UC), triglycerides (TG), phospholipids (PL), apolipoprotein A-I (apoA-I) and apolipoprotein B (apoB), will be determined periodically throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Connie Keyserling, MS, Study Director — Cerenis Therapeutics; Stephen Nicholls, MD PhD, Study Chair — South Australian Health and Medical Research Institute
Locations (35):
- United States (13):
  - Heart Center Research, LLC, Huntsville, Alabama
  - VA San Diego Healthcare System, San Diego, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - VA Eastern Colorado Health Care System, Denver, Colorado
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Cardiovascular Associates Research LLC, Covington, Louisiana
  - Cardiac and Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - University of Missouri Health System, Columbia, Missouri
  - Buffalo Heart Group LLP, Buffalo, New York
  - Veterans Affairs WNY Healthcare System, Buffalo, New York
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - South Oklahoma Heart Research, LLC, Oklahoma City, Oklahoma
  - Dallas VA Medical Center, Dallas, Texas
- Australia (8):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Queen Elizabeth Hospital, Woodville South, South Australia
  - Peninsula Heart Centre, Frankston, Victoria
  - Epworth Research Institute, Richmond, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Hungary (6):
  - Semmelweiss University, Budapest
  - Military Hospital, Budapest
  - University of Debrecen, Debrecen
  - Pándy Kálmán County Hospital, Gyula
  - County Hospital of Kecskemet, Kecskemét
  - University of Szeged, Szeged
- Netherlands (8):
  - Meander Medisch Centrum, Amersfoort
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Scheper Ziekenhuis, Emmen
  - Medisch Centrum Haaglanden, Leidschendam
  - Canisius-Wilhelmina hospital, Nijmegen
  - Maasstad Hospital, Rotterdam
  - Twee Steden hospital (Tilburg), Tilburg
  - VieCuri Medisch Centrum, Venlo

IPD SHARING:
Plan to Share IPD: Undecided
to be determined.

REFERENCES:
- [Derived] Nicholls SJ, Andrews J, Kastelein JJP, Merkely B, Nissen SE, Ray KK, Schwartz GG, Worthley SG, Keyserling C, Dasseux JL, Griffith L, Kim SW, Janssan A, Di Giovanni G, Pisaniello AD, Scherer DJ, Psaltis PJ, Butters J. Effect of Serial Infusions of CER-001, a Pre-beta High-Density Lipoprotein Mimetic, on Coronary Atherosclerosis in Patients Following Acute Coronary Syndromes in the CER-001 Atherosclerosis Regression Acute Coronary Syndrome Trial: A Randomized Clinical Trial. JAMA Cardiol. 2018 Sep 1;3(9):815-822. doi: 10.1001/jamacardio.2018.2121. PMID 30046828